CLINICAL TRIAL: NCT03832530
Title: Adherence to Periconception HIV Risk-reduction Among Uninfected Women in Rural Uganda
Brief Title: Periconception PrEP for HIV-exposed Ugandan Women
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Mbarara University of Science and Technology (Other)
Responsible Party: Principal Investigator, Lynn T Matthews, Principal Investigator, University of Alabama at Birmingham
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: 2017P001853
Record Dates: First submitted 2018-12-07; First posted 2019-02-06 (Actual); Last update posted 2021-05-26 (Actual); Status verified 2021-05

CONDITIONS: HIV Prevention
Keywords: PrEP; conception; prevention

STUDY DESIGN:
Intervention Model Description: Safer conception counseling
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: Yes

ARMS (1):
- HIV-uninfected women (Experimental): A sample of 150 women, aged 18-35, likely to be fertile based on reproductive health history, with reported personal or partner desire to have a child in the next year and who self-reports having a relationship with a partner she reports as HIV-infected or likely to be HIV-infected (e.g. taking medicine daily, goes to clinic routinely, has HIV-infected partners, he has implied that he is "sick" but has not disclosed). All women are offered comprehensive safe conception counseling -- this is the intervention -- inclusive of daily oral TDF/FTC as PrEP.
  Interventions: Behavioral: Safer conception counseling inclusive of periconception PrEP

INTERVENTIONS:
Behavioral: Safer conception counseling inclusive of periconception PrEP — Observational evaluation of factors associated with uptake of and adherence to daily, oral TDF/FTC PrEP and other safer conception methods (including: CHCT, ART for the infected partner, and uptake of contraception for those who decide not to conceive during follow-up) over 9 month. Maximum 19 month follow-up period (through pregnancy outcome).

SUMMARY:
In this mixed-methods research study, the study team will offer comprehensive safer conception services to 150 HIV-uninfected women reporting an HIV-infected or high-risk partner and personal or partner plans for pregnancy in rural Uganda to evaluate prevalence and determinants of uptake and adherence (tenofovir plasma concentration >40ng/mL, opening pill device to take >80% of dispensed pills) to PrEP and other safer conceptions strategies among Ugandan women exposed to HIV.

DETAILED DESCRIPTION:
The study plans to enroll 150 HIV-uninfected women with an HIV-positive or HIV-serostatus unknown partner and personal or partner pregnancy plans. Eligible women will participate in comprehensive safer conception counseling including offering daily, oral TDF/FTC as PrEP. The primary outcomes are to evaluate uptake of and adherence to periconception PrEP among HIV-exposed women in rural Uganda.

To accomplish this, women will participate in quarterly study visits, HIV and pregnancy testing, questionnaires and safer conception/adherence group counseling sessions. Participants will be eligible to initiate PrEP at any time during the first 6 months of the 9-month study follow-up period. Participants who initiate PrEP will use an electronic pill cap to measure daily adherence and will be asked to give blood samples to measure plasma TFV at quarterly study visits.

For women who become pregnant in the first 9 months, investigators will follow them up through completion of pregnancy to evaluate PrEP use, pregnancy and infant outcomes.

Study duration will be a maximum 19 month follow-up period (through pregnancy outcome) .

Investigators will offer objective sexually transmitted infection (STI) testing to all participants in order to measure the prevalence, incidence, and factors associated with STIs. Investigators will compare incidence among women who choose and who do not choose PrEP. Investigators will also measure the number of episodes of condomless sex each month as a mediator variable for STI development.

ELIGIBILITY:
Self Report Inclusion Criteria:

1. Female
2. Aged 18-35
3. Likely to be fertile based on reproductive health history [55]
4. Reported personal or partner desire to have a child in the next year [56-59]
5. With a partner she reports as HIV-infected or likely to be HIV-infected (e.g. taking medicine daily, goes to clinic routinely, has HIV-infected partners, he has implied that he is "sick" but has not disclosed).
6. Live within 60km of clinic. Not planning on relocating to an area incompatible with ability to attend quarterly clinic over a 9-month follow-up period

Objective Inclusion Criteria:

1. HIV-negative (onsite rapid testing)
2. Not currently pregnant (onsite urine b-hcg testing)
3. Fluent in English or local language
4. Otherwise able to participate in the informed consent process

Exclusion Criteria

1. Currently pregnant
2. HIV-positive

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes — Female
Enrollment: 150 (Actual)
Dates: Start 2017-11-27 (Actual); Primary Completion 2019-04-01 (Actual); Study Completion 2020-12-30 (Actual)

PRIMARY OUTCOMES:
Uptake of PrEP | 9 months
  Measure prevalence (measured by the proportion of women who collect the first 3 month supply of drug) TDF/FTC PrEP for safer conception

SECONDARY OUTCOMES:
Adherence to PrEP, daily pill taking behavior | 9 months
  We will measure the proportion of women who achieve daily adherence to at least 80% of PrEP through electronic pill count measurement
Adherence to PrEP, plasma levels | 9 months
  We will measure the proportion of women who achieve TFV plasma levels consistent with taking medication (detectable) and taking enough medication to confer protection (=>40ng/mL).

CONTACTS AND LOCATIONS:
Locations (1):
- Mbarara University of Science and Technology, Mbarara, Uganda

REFERENCES:
- [Derived] Matthews LT, Atukunda EC, Owembabazi M, Kalyebera KP, Psaros C, Chitneni P, Hendrix CW, Marzinke MA, Anderson PL, Isehunwa OO, Hurwitz KE, Bennett K, Muyindike W, Bangsberg DR, Haberer JE, Marrazzo JM, Bwana MB. High PrEP uptake and objective longitudinal adherence among HIV-exposed women with personal or partner plans for pregnancy in rural Uganda: A cohort study. PLoS Med. 2023 Feb 16;20(2):e1004088. doi: 10.1371/journal.pmed.1004088. eCollection 2023 Feb. PMID 36795763
- [Derived] Atukunda EC, Owembabazi M, Pratt MC, Psaros C, Muyindike W, Chitneni P, Bwana MB, Bangsberg D, Haberer JE, Marrazzo J, Matthews LT. A qualitative exploration to understand barriers and facilitators to daily oral PrEP uptake and sustained adherence among HIV-negative women planning for or with pregnancy in rural Southwestern Uganda. J Int AIDS Soc. 2022 Mar;25(3):e25894. doi: 10.1002/jia2.25894. PMID 35324081

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-05-03): https://cdn.clinicaltrials.gov/large-docs/30/NCT03832530/Prot_SAP_000.pdf